CLINICAL TRIAL: NCT05937932
Title: Inside Depression Clinical Trials: Patient Experiences Shared While Undergoing Clinical Trials
Brief Title: Exploring Clinical Study Experiences of People With Depression
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 82303651
Record Dates: First submitted 2023-06-30; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Depression
Keywords: depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study seeks to delve into the firsthand experiences of patients diagnosed with depression who partake in a separate clinical trial featuring a specific medical intervention. The primary emphasis will be on meticulously tracking the rates of trial completion and withdrawal among these individuals.

By joining this clinical trial, individuals have the unique opportunity to contribute to the betterment of future depression patients and play an active role in advancing medical research.

ELIGIBILITY:
Inclusion Criteria:

* Patient has self-identified as planning to enroll in a clinical trial
* Patient has been diagnosed with depression
* Patient is a minimum of 18 years or older

Exclusion Criteria:

* Patient does not understand, sign, and return consent form
* Inability to perform regular electronic reporting
* Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with depression who are actively considering enrolling in an observational clinical trial, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to participate in a depression clinical trial | 3 months
Rate of patients who remain in depression clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fancourt D, Steptoe A, Bu F. Trajectories of anxiety and depressive symptoms during enforced isolation due to COVID-19 in England: a longitudinal observational study. Lancet Psychiatry. 2021 Feb;8(2):141-149. doi: 10.1016/S2215-0366(20)30482-X. Epub 2020 Dec 9. PMID 33308420
- [Background] Dawson SR, Mallen CD, Gouldstone MB, Yarham R, Mansell G. The prevalence of anxiety and depression in people with age-related macular degeneration: a systematic review of observational study data. BMC Ophthalmol. 2014 Jun 12;14:78. doi: 10.1186/1471-2415-14-78. PMID 24923726
- [Background] Matison AP, Mather KA, Flood VM, Reppermund S. Associations between nutrition and the incidence of depression in middle-aged and older adults: A systematic review and meta-analysis of prospective observational population-based studies. Ageing Res Rev. 2021 Sep;70:101403. doi: 10.1016/j.arr.2021.101403. Epub 2021 Jul 8. PMID 34246793

DOCUMENTS (1):
  • Informed Consent Form (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT05937932/ICF_000.pdf